CLINICAL TRIAL: NCT03228108
Title: The Effect of Rectal Swab Culture-guided Antimicrobial Prophylaxis in Men Undergoing Prostate Biopsy on Infectious Complications and Cost of Care: A Randomized Controlled Trial in the Netherlands.
Brief Title: Culture-guided Antimicrobial Prophylaxis in Men Undergoing Prostate Biopsy.
Acronym: pro-SWAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: pro-SWAP104622
Record Dates: First submitted 2017-07-18; First posted 2017-07-24 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-11

CONDITIONS: Complication; Infection; Prostate Cancer
Keywords: Culture-guided; Targeted prophylaxis; Prostate biopsy; Antibiotic prophylaxis
MeSH Terms: conditions — Infections; Prostatic Neoplasms | interventions — Ciprofloxacin; Trimethoprim, Sulfamethoxazole Drug Combination; Fosfomycin; Amdinocillin Pivoxil; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted antimicrobial prophylaxis (Experimental): Men whose rectal swabs do not show ciprofloxacin-resistant bacteria will receive ciprofloxacin prior to biopsy (equal to the active comparator arm), and men whose swabs do show ciprofloxacin-resistant bacteria will receive alternative oral antibiotics, based on culture results, in the following order:
  * trimethoprim/sulfamethoxazole (SXT) 960 mg orally 2 hours before and 12 hours after prostate biopsy, or
  * fosfomycin 3 g orally 2 hours before prostate biopsy, or
  * pivmecillinam/augmentin respectively 400 mg and 500/125 mg 2 hours before prostate biopsy followed by 2 days with three divided doses each day after prostate biopsy.
  Interventions: Drug: Ciprofloxacin; Drug: Trimethoprim/Sulfamethoxazole; Drug: Fosfomycin; Drug: Pivmecillinam/augmentin
- Routine empirical prophylaxis (Active Comparator): Ciprofloxacin 500 mg orally 2 hours before and 12 hours after transrectal prostate biopsy.
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — see study arms.
  Other Names: Ciproxin
Drug: Trimethoprim/Sulfamethoxazole — see study arms.
  Other Names: Co-trimoxazole
  Arms: Targeted antimicrobial prophylaxis
Drug: Fosfomycin — see study arms.
  Other Names: Monuril
  Arms: Targeted antimicrobial prophylaxis
Drug: Pivmecillinam/augmentin — see study arms.
  Other Names: Selexid; Amoxicillin/clavulanic acid
  Arms: Targeted antimicrobial prophylaxis

SUMMARY:
This study aims to assess the effectiveness and cost-effectiveness of rectal swab culture-guided antimicrobial prophylaxis to reduce infectious complications after transrectal prostate biopsy. Half of participants will receive routine empirical prophylaxis with oral ciprofloxacin (control group), while the other half will receive rectal culture-guided oral antibiotic prophylaxis (intervention group). In the intervention group, men whose rectal swabs do not show ciprofloxacin-resistant bacteria will receive ciprofloxacin prophylaxis, comparable to the control group. In case of ciprofloxacin-resistant bacteria an alternative oral antibiotic based on the culture results will be prescribed (trimethoprim/sulfamethoxazole, fosfomycin or pivmecillinam/augmentin).

The investigators hypothesise that the targeted prophylaxis group (intervention group) will have a lower rate of post-biopsy infectious complications compared to the control group.

DETAILED DESCRIPTION:
Several classes of antibiotics are proven effective for prophylaxis during transrectal prostate biopsy, reducing infectious complications to less than 1% in case of susceptible rectal flora. Ciprofloxacin has been best studied and is recommended as first choice prophylaxis in urology guidelines. However, due to increasing fluoroquinolone resistance in gram negative bacilli (currently more than 20% in E.coli), a significant increase up to 6% in infectious complications after transrectal prostate biopsy was recently noticed. Antibiotic treatment of these infections and hospitalization may account for increased health care associated costs and will contribute to the further development of antibiotic resistance.

Besides, in urology guidelines no clear recommendations are made on the duration of prophylaxis. In the Netherlands, therefore, various prophylactic ciprofloxacin schedules are used, of which 2 to 3 day regimens are most common. Prolonged duration of prophylaxis during prostate biopsy is not proven to be more effective than a 1-day regimen, but it is more likely to select more fluoroquinolone (FQ) resistance.

This study aims to assess the effectiveness and cost-effectiveness of rectal culture-guided antimicrobial prophylaxis to reduce infectious complications after transrectal prostate biopsy. Also, duration of antibiotic prophylaxis will be minimized to 24 hours, thereby controlling further development of resistant bacteria.

The culture method used in this study with four phenotypic screening agars to support the choice of one of the oral prophylactic antibiotics is innovative. Culture results become available rapidly, within 48 hours, the method is simple, relatively inexpensive, as it does not need full susceptibility testing of separate colonies, and useful in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form.
* Subject undergoes a transrectal prostate biopsy as part of the standard care in the Radboudumc (Nijmegen), Canisius Wilhelmina hospital (Nijmegen) or Catharina hospital (Nijmegen) (because of suspicion of prostate cancer).

Exclusion Criteria:

* Inability to receive ciprofloxacin (e.g. documented history of sensitivity to medicinal products or excipients similar to those found in the antibiotic prophylaxis, relevant history or presence of cardiovascular disorders)
* Inability to receive either co-trimoxazole, fosfomycin and pivmecillinam/augmentin prophylaxis for any reason (e.g. documented history of sensitivity to medicinal products or excipients similar to those found in the antibiotic prophylaxis)
* Inability to understand the nature of the trial and the procedures required.
* Individuals with an urinary tract infection or acute prostatitis within 14 days prior to intervention.
* Individuals who receive antibiotics within 14 days before prostate biopsy.
* Individuals who fail to send a rectum swab to the microbiology laboratory.
* Individuals whose rectal swab shows no growth on a (growth) control MacConkey agar without antibiotics.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1538 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-09-26 (Actual)

PRIMARY OUTCOMES:
Any registered clinical infectious complication after prostate biopsy | within 7 days post-biopsy
  Urinary tract infection, pyelonephritis, sepsis, fever, acute prostatitis, acute epididymitis

SECONDARY OUTCOMES:
Cost of care | within 30 days after prostate biopsy
  Difference of costs between the intervention and the control group
Positive microbiological results | within 7 and 30 days after prostate biopsy
  Urine or blood culture results
Any registered clinical infectious complication after prostate biopsy | within 7 and 30 days after prostate biopsy
  Urinary tract infection, pyelonephritis, sepsis, fever, acute prostatitis, acute epididymitis
Hospitalization after prostate biopsy | within 30 days after prostate biopsy
  Any hospital admission, including ICU admission
Overall mortality | within 30 days after prostate biopsy
  Mortality of any cause
Side effects of used antibiotics | within 30 days after prostate biopsy
  All side effects mentioned in the Summary of Product Characteristics (SPC)
Prevalence of ciprofloxacin-resistant gram negative bacilli in local rectal flora | rectal swabs are taken 14 days before biopsy
  Assessed through microbiological rectal swab cultures
Overall antibiotic use after prostate biopsy | within 30 days after prostate biopsy
  Number of antibiotic prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Heiman Wertheim, Prof. dr., Study Director — Radboud University Medical Center
Locations (13):
- Netherlands (13):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Rijnstate, Arnhem
  - Bravis, Bergen op Zoom
  - Amphia Hospital, Breda
  - Catharina Hospital, Eindhoven
  - Zuyderland Hospital, Heerlen
  - Canisius Wilhelmina Hospital, Nijmegen
  - Radboud University Medical Center, Nijmegen
  - Bravis, Roosendaal
  - Zuyderland Hospital, Sittard
  - Elisabeth Tweesteden Hospital, Tilburg
  - Bernhoven Hospital, Uden
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tops SCM, Kolwijck E, Koldewijn EL, Somford DM, Delaere FJM, van Leeuwen MA, Breeuwsma AJ, de Vocht TF, Broos HJHP, Schipper RA, Steffens MG, Wegdam-Blans MCA, de Brauwer E, van den Bijllaardt W, Leenders ACAP, Sedelaar JPM, Wertheim HFL, Adang E. Cost Effectiveness of Rectal Culture-based Antibiotic Prophylaxis in Transrectal Prostate Biopsy: The Results from a Randomized, Nonblinded, Multicenter Trial. Eur Urol Open Sci. 2023 Feb 26;50:70-77. doi: 10.1016/j.euros.2023.02.006. eCollection 2023 Apr. PMID 37101774
- [Derived] Tops SCM, Kolwijck E, Koldewijn EL, Somford DM, Delaere FJM, van Leeuwen MA, Breeuwsma AJ, de Vocht TF, Broos HJHP, Schipper RA, Steffens MG, Teerenstra S, Wegdam-Blans MCA, de Brauwer E, van den Bijllaardt W, Leenders ACAP, Sedelaar JPM, Wertheim HFL. Rectal Culture-Based Versus Empirical Antibiotic Prophylaxis to Prevent Infectious Complications in Men Undergoing Transrectal Prostate Biopsy: A Randomized, Nonblinded Multicenter Trial. Clin Infect Dis. 2023 Apr 3;76(7):1188-1196. doi: 10.1093/cid/ciac913. PMID 36419331